CLINICAL TRIAL: NCT07014098
Title: Effectiveness of Robot-Aided Off-Axis Neuromuscular Training for Knee Osteoarthritis: A Randomized Controlled Trial
Brief Title: Robot-Aided Off-Axis Neuromuscular Training for Knee OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Li-Qun Zhang, Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HP-00113883
Record Dates: First submitted 2025-04-25; First posted 2025-06-10 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis of Knee
Keywords: knee osteoarthritis; robot-assisted; neuromuscular training; knee biomechanics; knee symptoms; evaluation-based training strategy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- evaluation-based, progressive, off-axis neuromuscular training group (Experimental)
  Interventions: Device: Robot-Aided Off-Axis Neuromuscular Training
- traditional elliptical regular stepping group (Sham Comparator)
  Interventions: Device: Traditional elliptical regular stepping

INTERVENTIONS:
Device: Robot-Aided Off-Axis Neuromuscular Training — A novel custom-designed elliptical trainer is developed, and its footplates are robot-controlled to be moved in four off-axis directions (sliding in/out, pivoting in/out; corresponding to knee valgus/varus, internal rotation/external rotation). Before the training, off-axis neuromechanical assessments will be conducted to determine which specific off-axis direction (valgus, varus, internal rotation, external rotation, or combination of the off-axis directions) has neuromechanical deficits. During the evaluation-based and subject-specific neuromuscular training, the different training modes will be conducted progressively from regular stepping, footplate position control, spring mode, perturbation, to slippery mode.
  Arms: evaluation-based, progressive, off-axis neuromuscular training group
Device: Traditional elliptical regular stepping — traditional elliptical regular stepping
  Arms: traditional elliptical regular stepping group

SUMMARY:
Although the primary knee motion occurs in flexion/extension, the frontal and transverse (off-axis) knee motions are smaller but crucial for maintaining joint stability and normal knee loading. Altered kinematics and neuromuscular control in off-axis knee motions have been reported in patients with knee osteoarthritis (OA), which are associated with excessive knee loading and the progression of knee OA. However, traditional rehabilitative treatments for people with knee OA and existing exercise equipment often focus on sagittal plane movement. Probably due to the technical limitations, there is a lack of convenient and effective equipment/method to train patients with knee OA in off-axis (frontal and transverse) planes.

The purpose of this study is to use a robot-aided elliptical training device to measure knee neuromechanical properties and to improve neuromuscular control in off-axis knee motions, aiming for joint de-loading and pain reduction for individuals with knee OA.

DETAILED DESCRIPTION:
The device used in this study is provided by Rehabtek LLC, which has received U.S. federal grants to develop and commercialize this device.

Eligible knee osteoarthritis (OA) patients will be randomly assigned to three groups: (A) evaluation-based, progressive, neuromuscular training group; (B) traditional regular stepping group.

Participants in both groups will undergo 3 assessments.

Once the participants have consented, the first assessment visit will be scheduled before the training, which includes the neuromechanical and clinical assessments:

1. The neuromechanical assessments involve the off-axis knee moments and instability during the free-speed stepping and fast stepping tasks on the elliptical machine to see which off-axis directions (knee valgus, varus, internal rotation, and/or external rotation) or combination of directions show excessive moments. Off-axis instability, muscle strength, range of motion, stiffness, proprioception acuity, and knee moments during stepping will also be evaluated.

   A. Knee frontal-plane neuromechanical properties.
   * The participants sit with their knees in 0 degrees flexion. A fixture is used to hold the thigh near the femoral condyles steadily. The footplate is moved by a linear motor mediolaterally in the frontal plane, a 6-axis force sensor underneath the footplate, and a 6-DOF(degree of freedom) goniometer on the knee is used to measure knee motions. With the knee joint perturbed in varus-valgus motion, varus-valgus angle and torque can be determined.
   * With the participants in the seated position and relaxed, the participants' knee varus-valgus laxity and passive range of motion (ROM) will be determined when a specific passive resistance torque is reached at varus or valgus direction.
   * Knee varus-valgus proprioceptive acuity is measured by the threshold to detection of a passive movement in the respective varus and valgus directions. From the neutral position, the knee is randomly moved into either varus or valgus direction by the linear motor at a constant, slow speed. The blindfolded participant is instructed to push a trigger and report the direction of motion when he/she first sense which direction the knee is moving into. The motor stops the movement once the trigger is activated. Each participant completes 8 trials without complaints of pain or discomfort.
   * Tibial varus-valgus pain threshold is measured by the threshold to feel pain in the respective tibial varus-valgus directions. While the participant is seated relaxed, the footplate moves in varus-valgus direction. This movement occurs at a constant speed. The participant is asked to push a trigger and report the direction of pain when he/she first senses and the motor would stop and move back to the initial position.
   * For the active muscular contribution to varus-valgus stiffness, with the subject seated at 0 deg knee flexion, participants' ability to actively stabilize the lower leg against perturbations in varus-valgus direction is evaluated. First, the participants are relaxed and in a seated position while the footplate moves medially and laterally until a specific resistance torque limit is reached in each direction. Second, the participant is asked to resist medial-lateral movements imposed by the footplate. Active muscular contribution to varus-valgus stiffness is determined as the difference in stiffness between these two conditions.
   * Muscle strength measurement in varus-valgus direction With the subject seated at 0-degree knee flexion, the researchers examine the ability of the participants to actively generate torque in the frontal plane. The footplate is locked in the neutral position. Then the subject is asked to perform maximal voluntary isometric contraction in varus direction against the footplate. The participants are provided with real-time visual feedback of the amount of torque they generate. Then, the participants are asked to hold the maximum contraction for 4 seconds and then release it. The task is performed 3 times. Then, the participants are given 30 seconds of rest between each trial.

   The same procedure will be repeated for the evaluation of their valgus torque generation ability.

   B. Tibial internal-external rotation neuromechanical properties
   * Knee axial plane neuromechanical properties are quantified with the leg axially rotated by a pivoting motor underneath the footplate. Considering that femoral rotation is coupled with tibial rotation at extended knee positions, the test is conducted in the seated position, and the knee is flexed at 90 degrees to minimize the coupled rotations and allow for reliable testing of tibial rotation relative to the femur. The foot is strapped to the footplate with a 6-axis force sensor underneath. The tibial long axis is aligned with the Z-axis of the 6-axis force sensor and the pivoting motor underneath.
   * The zero tibial rotation angle is set with the second toe directed forward. To determine the torque-rotation relationship and joint ROM in tibial internal and external rotation, the foot and tibia are rotated slowly by the pivoting servomotor until a preset resistance torque (or position) limit is reached. The driving device then stops for 2 seconds before reversing the movement direction and rotating the knee until the preset torque (or position) limit in the opposite direction is reached. The position limits are determined manually by rotating the subject's tibia to the extreme internal and external rotation positions (within comfortable limits for the subject). Joint torque and force are measured continuously using the 6-axis torque sensor. Motor rotation is measured continuously using the motor encoder, and the 6-DOF goniometer is used to measure the knee motion directly.
   * Tibial internal-external rotation proprioceptive acuity is measured by the threshold to detection of a passive movement in the respective tibial internal or external rotation directions. From the neutral position, the knee is randomly moved into either tibial internal or external rotation direction by the pivoting motor at a constant, slow speed. The participant is instructed to push a trigger and report the direction of motion when he/she first sense which direction the knee is moving into. The motor stops the movement once the trigger is activated. Each participant completes 8 trials without complaints of pain or discomfort. Proprioceptive acuity is quantified by the tibial internal-external rotation angle, where the participant senses the motion, with a greater angle indicating worse acuity.
   * Tibial Internal-External Rotation Pain Threshold Tibial internal-external rotation pain threshold is measured by the threshold to feel pain in the respective tibial internal or external rotation directions. While the participant is seated relaxed, the footplate rotates in internal or external rotation direction, which induces tibial rotations. This movement occurs at a constant speed. The participant is asked to push a trigger and report the direction of pain when he/she first senses and the motor would stop and move back to the initial position.
   * Active muscular contribution to tibial internal-external rotation stiffness With the subject seated at 90 ° knee flexion, the researchers examine the ability of the subject to actively stabilize the lower leg against perturbations in directions of tibial internal/external rotations. First, the subject's seat relaxed while the footplate rotates internally and externally until a specific resistance torque limit is reached. Second, the participant is asked to resist the internal/external rotations imposed by the footplate. Active muscular contribution to tibial internal/external rotation stiffness is determined as the difference in stiffness between these two conditions.
   * Muscle strength measurement in producing internal/external rotation torque With the subject seated at 90-degree knee flexion, the ability of the subject to actively generate internal/external rotation torque is assessed. The footplate is locked in the neutral position. Then, the subject is asked to perform maximal voluntary isometric contraction of internal rotation against the footplate. The participants are provided with real-time visual feedback of the amount of torque they generate. Then, the participants are asked to hold the maximum contraction for 4 seconds and then release it. The participants perform the task 3 times. Then, the participants are given 30 seconds of rest between each trial.

   The same procedure will be repeated for the evaluation of participants' external rotation torque generation ability.

   C. Tests of walking

   - To evaluate participant gait biomechanics, a motion capture system is employed for recording overground walking behavior over a short distance with markers attached to the lower limbs, upper limbs, and trunk. This assessment is performed in the first evaluation session and during the following assessment sessions.

   D. Dynamic structural changes

   - The SWEU (Aixplorer Version 4.2; Supersonic Imagine, Aix-en-Provence, France) will be synchronized with the robot-controlled elliptical device. The ultrasound probe (4-15 MHz, Super Liner 15-4; Supersonic Imagine) will be stabilized by a 3-D printed holder at the medial knee to make sure the distal femur and proximal tibia can be visualized. The stiffness of distal femur and proximal tibia cartilage, and meniscus extrusion will be calculated at each time point that corresponds to the pain and stiffness test in the 4 off-axis knee motions.
2. The subject will be asked to complete self-reported outcome measure, including the knee injury and osteoarthritis outcome score (KOOS) or international knee documentation committee (IKDC), the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), SF-36, the Fremantle Knee Awareness Questionnaire (FreKAQ), Rated Perceived Exertion (RPE) Scale, Tegner activity scale, and visual analogue scale (VAS). The subjects also perform the Four Square Step Test, the 6-minute walk test, the 20-meter walk test, and time up and go (TUG), the 30-second sit-to-stand test. The passive and active range of motion of lower limb joints will be assessed. These evaluations are part of the clinical assessment. Knee girth and Q-angle will be measured as well. Single-leg squat and single-leg hop tests may be used as well.

The subjects will do off-axis training on the elliptical stepping system in our lab. The elliptical stepping system can detect the forces and torques in the lower limb during free-speed stepping and fast stepping and give real-time visual feedback if forces in one direction are excessive.

Training in group A will be based on the specific biomechanical needs of each subject. We will put the footplates of the elliptical in specific outward/inward positions or make some modifications to the foot position in the sagittal and frontal planes. Then the researchers ask subjects to perform stepping on the elliptical at their self-selected speed. Training in group B will be traditional elliptical regular stepping.

For both group A & B, the training protocol will be conducted 3 times a week for 5 weeks. Each training session will last about 40 minutes. The amount of usual care in all three groups will be documented and considered as a potential cofounder in the statistical analysis.

For groups A & B, after the 5-week training ends, the same outcome measures will be reassessed immediately after the training, and 8 weeks post-training as the initial visit.

Healthy age-sex matched subjects undergo one assessment session. All the assessment procedures mentioned above will be conducted for healthy subjects as well, except the pain threshold detection section and self-reported outcome measures (KOOS, IKDC, WOMAC, and VAS).

As part of the assessment and training sessions, the researchers will measure participants' blood pressure, heart rate, and oxygen saturation level at the beginning and the end of each session. The researchers will also monitor participants' heart rate and oxygen saturation during the elliptical test.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 - 85 years.
* Meets the ACR classification criteria for knee OA (clinical + radiographic criteria); Kellgren-Lawrence grade I-III.
* Persistent knee pain ≥ 3 months.
* Able to independently complete elliptical training (6 minutes without interruption).

Exclusion Criteria:

* Other inflammatory joint diseases (e.g., rheumatoid arthritis).
* Knee trauma, surgery, or intra-articular injections within the past year.
* History of knee or hip replacement.
* Cardiovascular disease or uncontrolled hypertension contradict to exercises.
* Cognitive impairment (Montreal cognitive assessment < 22).
* Currently participating in another interventional study for the lower limb.
* Neurological impairment (e.g., stroke, Parkinson's disease, radicular pain).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Peak knee adduction moment | Baseline, immediately after the 5-week training, and follow-up evaluation 8-week post-training
Knee pain | Baseline, immediately after the 5-week training, and follow-up evaluation 8-week post-training
  Questionnaires, including the Knee Injury and Osteoarthritis Outcome Score (KOOS)

SECONDARY OUTCOMES:
Knee proprioception acuity/pain in off-axis directions | Baseline, immediately after the 5-week training, and follow-up evaluation 8-week post-training
Knee range of motions/stiffness/laxity in off-axis directions | Baseline, immediately after the 5-week training, and follow-up evaluation 8-week post-training
Functional ability | Baseline, immediately after the 5-week training, and follow-up evaluation 8-week post-training
  Time-up-and-go test (usual and fast speed) and 6-minute walking test
Heath-related quality of life | Baseline, immediately after the 5-week training, and follow-up evaluation 8-week post-training
  Assessed by the SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Qun Zhang, PhD, Principal Investigator — University of Maryland, Baltimore

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant-level data (demographics, outcomes, lab results, etc.); study documents, such as protocols, statistical analysis plans, and case report forms; and clinical study reports (CSRs) with anonymized results.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The IPD and supporting information will be available from Oct 2025, for 5 years.
Access Criteria: Who: Researchers (academic, clinical, or industry) who provide a methodologically sound proposal for approved scientific use. Regulatory authorities (e.g., FDA, EMA) for review and compliance verification. Ethics committees or auditors for validation of study integrity.
  What: De-identified participant-level data (demographics, outcomes, lab results, etc.). Study documents, such as protocols, statistical analysis plans, and case report forms. Clinical study reports (CSRs) with anonymized results.
  How: Researchers must submit a formal proposal to a designated data-sharing platform (e.g., ClinicalStudyDataRequest.com) or the study sponsor. Approved requesters sign a data use agreement (DUA) and receive secure access via encrypted repositories or controlled cloud-based platforms.

REFERENCES:
- [Background] Lee SJ, Ren Y, Geiger F, Chang AH, Press JM, Zhang LQ. Offaxis neuromuscular training of knee injuries using an offaxis robotic elliptical trainer. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:2081-4. doi: 10.1109/IEMBS.2011.6090386. PMID 22254747
- [Background] Griffin LY, Agel J, Albohm MJ, Arendt EA, Dick RW, Garrett WE, Garrick JG, Hewett TE, Huston L, Ireland ML, Johnson RJ, Kibler WB, Lephart S, Lewis JL, Lindenfeld TN, Mandelbaum BR, Marchak P, Teitz CC, Wojtys EM. Noncontact anterior cruciate ligament injuries: risk factors and prevention strategies. J Am Acad Orthop Surg. 2000 May-Jun;8(3):141-50. doi: 10.5435/00124635-200005000-00001. PMID 10874221
- [Background] Williams GN, Chmielewski T, Rudolph K, Buchanan TS, Snyder-Mackler L. Dynamic knee stability: current theory and implications for clinicians and scientists. J Orthop Sports Phys Ther. 2001 Oct;31(10):546-66. doi: 10.2519/jospt.2001.31.10.546. PMID 11665743
- [Background] Ren Y, Lee SJ, Park HS, Zhang LQ. A pivoting elliptical training system for improving pivoting neuromuscular control and rehabilitating musculoskeletal injuries. IEEE Trans Neural Syst Rehabil Eng. 2013 Sep;21(5):860-8. doi: 10.1109/TNSRE.2013.2273874. PMID 24013591
- [Background] Lee SJ, Ren Y, Geiger F, Zhang LQ. Gender differences in offaxis neuromuscular control during stepping under a slippery condition. Eur J Appl Physiol. 2013 Nov;113(11):2857-66. doi: 10.1007/s00421-013-2727-3. Epub 2013 Sep 24. PMID 24062010
- [Background] Kang SH, Lee SJ, Ren Y, Zhang LQ. Real-time knee adduction moment feedback training using an elliptical trainer. IEEE Trans Neural Syst Rehabil Eng. 2014 Mar;22(2):334-43. doi: 10.1109/TNSRE.2013.2291203. PMID 24608687
- [Background] Tsai LC, Lee SJ, Yang AJ, Ren Y, Press JM, Zhang LQ. Effects of Off-Axis Elliptical Training on Reducing Pain and Improving Knee Function in Individuals With Patellofemoral Pain. Clin J Sport Med. 2015 Nov;25(6):487-93. doi: 10.1097/JSM.0000000000000164. PMID 25591131
- [Background] Lin CY, Tsai LC, Press J, Ren Y, Chung SG, Zhang LQ. Lower-Limb Muscle-Activation Patterns During Off-Axis Elliptical Compared With Conventional Gluteal-Muscle-Strengthening Exercises. J Sport Rehabil. 2016 May;25(2):164-72. doi: 10.1123/jsr.2014-0307. Epub 2015 May 6. PMID 25946669
- [Background] Lee SJ, Ren Y, Press JM, Lee J, Zhang LQ. Improvement in Offaxis Neuromuscular Control Under Slippery Conditions Following Six-Week Pivoting Leg Neuromuscular Training. IEEE Trans Neural Syst Rehabil Eng. 2017 Nov;25(11):2084-2093. doi: 10.1109/TNSRE.2017.2705664. Epub 2017 May 18. PMID 28541212
- [Background] Lauder TD, Baker SP, Smith GS, Lincoln AE. Sports and physical training injury hospitalizations in the army. Am J Prev Med. 2000 Apr;18(3 Suppl):118-28. doi: 10.1016/s0749-3797(99)00174-9. PMID 10736548
- [Background] Hootman JM, Dick R, Agel J. Epidemiology of collegiate injuries for 15 sports: summary and recommendations for injury prevention initiatives. J Athl Train. 2007 Apr-Jun;42(2):311-9. PMID 17710181